CLINICAL TRIAL: NCT04719208
Title: Reduction of Sars-CoV-2 Oral Viral Load With Prophylactic Mouth Rinse
Brief Title: [COVID-19] Reduction of Sars-CoV-2 Oral Viral Load With Prophylactic Mouth Rinse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ryan F. Bloomquist, Assistant Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: [1607808
Record Dates: First submitted 2020-10-21; First posted 2021-01-22 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Water; Mouthwashes; chlorhexidine gluconate; Hydrogen Peroxide; Povidone-Iodine; Ethanol; Listerine; Fumigant 93

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Chlorhexidine gluconate (A) (Experimental): Mouth rinse with 0.2% Chlorhexidine gluconate,
  Interventions: Other: Chlorhexidine gluconate (A) Mouth rinse with the solution provided
- Hydrogen peroxide (B) (Experimental): Mouth rinse with 1.5% hydrogen peroxide
  Interventions: Other: Hydrogen peroxide (B) Mouth rinse with the solution provided
- Betadine (C) (Experimental): Mouth rinse with betadine mouthwash,
  Interventions: Other: Betadine (C) Mouth rinse with the solution provided
- Mouth wash (D) (Experimental): Mouth rinse with alcohol-based mouthwash
  Interventions: Other: Alcohol mouthwash (Listerine) (D) Mouth rinse with the solution provided
- Water (E) (Placebo Comparator): Mouth rinse with water
  Interventions: Other: Water (E) Mouth rinse with the solution provided

INTERVENTIONS:
Other: Water (E) Mouth rinse with the solution provided — Subject will be asked to perform a simple mouth rinse for 2 minutes with one of the 5 mouth washes to be tested.
  Arms: Water (E)
Other: Chlorhexidine gluconate (A) Mouth rinse with the solution provided — Subject will be asked to perform a simple mouth rinse for 2 minutes with one of the 5 mouth washes to be tested.
  Arms: Chlorhexidine gluconate (A)
Other: Hydrogen peroxide (B) Mouth rinse with the solution provided — Subject will be asked to perform a simple mouth rinse for 2 minutes with one of the 5 mouth washes to be tested.
  Arms: Hydrogen peroxide (B)
Other: Betadine (C) Mouth rinse with the solution provided — Subject will be asked to perform a simple mouth rinse for 2 minutes with one of the 5 mouth washes to be tested.
  Arms: Betadine (C)
Other: Alcohol mouthwash (Listerine) (D) Mouth rinse with the solution provided — Subject will be asked to perform a simple mouth rinse for 2 minutes with one of the 5 mouth washes to be tested.
  Arms: Mouth wash (D)

SUMMARY:
The purpose of this study is to test the effectiveness of prophylactic mouth rinses in reducing the amount of viruses, specifically SARS-CoV-2 in the oral cavity. This research will guide dental and medical providers on best practices to be performed prior to dental and medical procedures involving the oral cavity.

DETAILED DESCRIPTION:
In response to SARS-CoV-2 the dental and greater healthcare communities have devised ways to combat the spread of the virus. Many dentists and physicians have advocated the use of prophylactic oral rinses for reduction of COVID-19 viral load in all patients prior to treatment in the oral pharyngeal cavity, but the effectiveness of these measures has not been validated with empirical evidence. The investigators will test COVID-19 positive hospital inpatients before and after the use of different combinations of oral rinses to provide guidance on best measures for dental or medical treatment. This research is imperative and essential as prophylactic rinses are already being used at AU and globally, without data to support their effectiveness specifically in COVID-19 positive patients.

Oral rinses have been used as an industry standard in dentistry for decades to reduce oral levels of pathogens including bacteria and viruses. According to the American Academy of Dentistry mouth rinses can be broken down into two categories, cosmetic and therapeutic. Those categorized as therapeutic include chlorhexidine, essential oils, fluoride, and hydrogen peroxide. These rinses are routinely used in both dental practices as well as in the OR setting prior to any invasive procedure involving treatment of the oral cavity. However, these mouth rinses, are typically utilized to reduce risk of infection to the patient. By disinfecting the oral cavity through bacteriostatic, bactericidal, and virucidal rinses practitioners can mitigate the risk of spreading an infection from a patient's mouth or the outside environment to other parts of their body. Prophylactic rinses are often used prior to routine dental procedures like fillings and cleaning to more invasive interventions like jaw reconstruction and tumor resection. This simple, cheap and innocuous procedure is now being used for a different purpose. In light of the COVID-19 pandemic, reduction in the spread of oral and respiratory borne viruses has become paramount in the global battle against coronavirus. Both dentists and medical providers, including ear nose throat specialists and anesthesiologists who routinely intubate patients, have implemented the use of these virucidal mouth rinses to reduce viral loads of both COVID-19 positive and non-infected patients. Dentists are particularly at risk for transmission of COVID-19 because they work directly in the oral cavity where the virus resides and the work they do creates an enormous amount of aerosols. In addition to a multitude of barrier and personal protective equipment (PPE) techniques being implemented, prior to procedures in the oral cavity patients are asked to rinse and spit different regimens of mouth rinses to reduce the chance of spreading SARS-CoV-2 to healthcare staff.

While healthcare workers have had to act quickly to respond to the pandemic and reduce the risk of spreading coronavirus, there is a lack of empirical evidence to support current practices. Here the investigators aim to address three questions; 1: Does oral prophylaxis effectively reduce oral viral load specifically of SARS-CoV-2; 2: If so for what duration is oral prophylaxis effective before viral load recovers in the oral cavity; 3: Which combination of virucidal prophylaxis if any is most effective.

ELIGIBILITY:
Inclusion Criteria:

1. Subject of both sexes, aged 18 years or older
2. Patients who are confirmed positive for COVID-19.
3. Patients currently hospitalized at Augusta University Medical Center.
4. Subject voluntarily signing the informed consent document.

Exclusion Criteria:

1. Age younger than 18 years old.
2. Patients that are tested negative for COVID-19
3. Patient who are intubated or too sick to give consent for the study.
4. Not able to speak in English or illiterate or lacking the decision-making capacity to consent for study.
5. Known allergy to Listerine, Betadine or Chlorhexidine gluconate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in oral SARS-CoV-2 load in oral cavity of COVID-19 patient using prophylactic mouth rinse | up to 2 hours post-rinse with mouthwash.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Augusta University, Augusta, Georgia
  - Augusta University-Dental College of Georgia, Augusta, Georgia

IPD SHARING:
Plan to Share IPD: No